CLINICAL TRIAL: NCT00003325
Title: Intraoperative Lymphatic Mapping in Patients With Stage I and II Squamous Carcinoma of the Vulva
Brief Title: Lymphatic Mapping in Treating Patients With Stage I or Stage II Cancer of the Vulva
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0173; CDR0000066277 (Other: CDR); NCI-2009-00579 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Vulvar Cancer
Keywords: stage I vulvar cancer; stage II vulvar cancer; squamous cell carcinoma of the vulva
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sentinenal lymph node mapping (Other): Sentinenal lymph node mapping
  Interventions: Procedure: Sentinel lymph node mapping

INTERVENTIONS:
Procedure: Sentinel lymph node mapping — Sentinel lymph node mapping

SUMMARY:
RATIONALE: Lymphatic mapping may improve the ability to detect cancer of the vulva.

PURPOSE: This phase III trial is studying how well lymphatic mapping works in treating patients with stage I or stage II cancer of the vulva.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the negative predictive value of a negative sentinel lymph node in patients with invasive squamous cell carcinoma of the vulva.
* Determine the location of the sentinel node in these patients.

OUTLINE: Patients receive injection(s) of isosulfan blue into the dermis at the junction of the tumor and normal vulvar skin. Once the afferent lymphatic channel and sentinel node have been identified, patients undergo unilateral or bilateral inguinal-femoral lymphadenectomy followed by resection of the primary tumor with adequate margins. Preoperative lymphoscintigraphy is also performed.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter or until recurrence.

PROJECTED ACCRUAL: A total of 40-630 patients will be accrued for this study within 2-6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive squamous cell carcinoma of the vulva that is greater than 1 mm in thickness as measured from the nearest rete peg

  * Tumor size must be 2-6 cm
  * No recurrent disease
* Prior excision of the primary disease or a history of carcinoma in situ of the vulva allowed
* No tumor extending into the urethra, anus, vagina, rectum, or bladder
* No grossly suspicious or inflamed groin nodes on physical exam
* No grossly infected primary tumors

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* GOG 0-3

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other invasive malignancy within the past 5 years except non-melanomatous skin cancer
* No known hypersensitivity to phenylethane compounds

PRIOR CONCURRENT THERAPY:

* No prior cancer therapy that contraindicates therapy in this study

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics
* No prior groin dissection

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 1999-12; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Predictive value of negative sentinel lymph nodes in vulvar cancer patients | at time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Charles Levenback, MD, Study Chair — M.D. Anderson Cancer Center
Locations (72):
- United States (72):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Todd Cancer Institute at Long Beach Memorial Medical Center, Long Beach, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Gynecologic Oncology of Indiana, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Maine Medical Center - Bramhall Campus, Portland, Maine
  - Harry & Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Women's Cancer Center - Lake Mead, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Saint Francis Campus, Tulsa, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Baptist Centers for Cancer Care, Memphis, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern University Hospital - Zale Lipshy, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - LDS Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Carilion Gynecologic Oncology Associates, Roanoke, Virginia
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin

REFERENCES:
- [Result] Levenback CF, Ali S, Coleman RL, Gold MA, Fowler JM, Judson PL, Bell MC, De Geest K, Spirtos NM, Potkul RK, Leitao MM Jr, Bakkum-Gamez JN, Rossi EC, Lentz SS, Burke JJ 2nd, Van Le L, Trimble CL. Lymphatic mapping and sentinel lymph node biopsy in women with squamous cell carcinoma of the vulva: a gynecologic oncology group study. J Clin Oncol. 2012 Nov 1;30(31):3786-91. doi: 10.1200/JCO.2011.41.2528. Epub 2012 Jul 2. PMID 22753905
- [Result] Levenback CF, Tian C, Coleman RL, et al.: Sentinel node (SN) biopsy in patients with vulvar cancer: A Gynecologic Oncology Group (GOG) study. [Abstract] J Clin Oncol 27 (Suppl 15): A-5505, 2009.